CLINICAL TRIAL: NCT02436148
Title: Reliability and Validity of the Finnish Version of the Prothesis Evaluation Questionnaire
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Jussi Repo, Researcher, Helsinki University Central Hospital
Other Study IDs: 364/13/03/02/2014/1
Record Dates: First submitted 2015-05-02; First posted 2015-05-06 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Amputation Stump
Keywords: PEQ validation study, Finland

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Prosthetic for major lower limb amputation — Prosthetic for major lower limb amputee

SUMMARY:
The present study assesses the reliability and validity of the Finnish version of Prothesis Evaluation Questionnaire. Major lower extremity amputees who use prosthesis are requited for the present study from the Helsinki and Uusimaa Hospital District and the Central Finland Health Care District.

DETAILED DESCRIPTION:
> 100 lower extremity prosthetic users with major lower extremity amputation are recruited for the present study. The aim is to assess the reliability and validity of the Finnish version of the Prothesis Evaluation Questionnaire (PEQ). The participants fill in a pre information form, the PEQ, the 15D health-related quality of life questionnaire, Houghton prothesis questionnaire, Locomotor Capabilities Index - 5, Prothesis Evaluation Questionnaire Mobility Section - 5. The psychometric abilities of the PEQ instrument are analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Major lower extremity amputation Prothetization

Exclusion Criteria:

* Other amputation besides major lower extremity
* No prothesis in use

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with major lower extremity amputation who has been prothetized.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Assessing the reliability and validity of the PEQ questionnaire | 1-10 years

SECONDARY OUTCOMES:
Prothesis Evaluation Questionnaire | 1-10 years
Houghton prothesis user score | 1-10 years
Locomotor Capabilities Index - 5 | 1-10 years
Prothesis Evaluation Questionnaire Mobility Section - 5 | 1-10 years

CONTACTS AND LOCATIONS:
Overall Officials: Erkki J Tukiainen, MD,PhD, Study Director — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki, Uusimaa
  - Central Finland Central Hospital, Jyväskylä